CLINICAL TRIAL: NCT04384367
Title: A Multicenter, Double-blind, Double-dummy, Randomized, Single-dose, Placebo-controlled Study to Evaluate the Efficacy and Safety of Rizatriptan-Naproxen (10/550 Mg) in the Acute Treatment of Migraine
Brief Title: Efficacy and Safety of Rizatriptan-Naproxen (10/550 Mg) in the Acute Treatment of Migraine
Acronym: RELIEF
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eurofarma Laboratorios S.A. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: EF167
Record Dates: First submitted 2020-04-06; First posted 2020-05-12 (Actual); Last update posted 2025-02-14 (Actual); Status verified 2025-02

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — rizatriptan; Naproxen; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Rizatriptan 10mg+ Naproxen 550mg (Experimental): Rizatriptan 10mg+ Naproxen 550mg
  Interventions: Drug: Rizatriptan 10 mg + Naproxen 550mg
- Maxalt 10mg (Active Comparator): Rizatriptan10mg
  Interventions: Drug: Maxalt 10Mg Tablet
- Flanax 550mg (Active Comparator): Naproxen 550mg
  Interventions: Drug: Flanax 550mg
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo oral tablet

INTERVENTIONS:
Drug: Rizatriptan 10 mg + Naproxen 550mg — oral - single dose
  Other Names: Medicamento
  Arms: Rizatriptan 10mg+ Naproxen 550mg
Drug: Maxalt 10Mg Tablet — oral - single dose
  Other Names: Medicamento
  Arms: Maxalt 10mg
Drug: Flanax 550mg — oral - single dose
  Other Names: Medicamento
  Arms: Flanax 550mg
Drug: Placebo oral tablet — oral - single dose
  Other Names: Medicamento
  Arms: Placebo

SUMMARY:
A phase III study, multicenter, double-blind, double-dummy, randomized, single-dose, placebo-controlled study to evaluate the efficacy and safety of Rizatriptan-Naproxen (10/550 mg) in the acute treatment of migraine.

⚠️Study will only be conducted in research centers in Brazil (please do not send e-mail if your center is outside brazil).

DETAILED DESCRIPTION:
This is a prospective, randomized, double-blind, double-dummy and placebo-controlled study in individuals with disabling migraine. The participants will be randomized to receive Rizatriptan + Naproxen (10/550mg), Rizatriptan (10mg), Naproxen (550mg) or placebo.

⚠️Study will only be conducted in research centers in Brazil (please do not send e-mail if your center is outside brazil).

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes;
* Aged between 18 and 65 years old;
* Capable and willing to give free and informed informed consent in writing;
* Migraine patients with or without aura, according to the International Headache Society (IHS).

Exclusion Criteria:

* Chronic migraine;
* Headache other than migraine (that is, tension-type headache, sinusitis, etc.).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2068 (Actual)
Dates: Start 2022-12-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-30 (Actual)

PRIMARY OUTCOMES:
2-hour pain-free | 11 weeks
  2-hour pain-free response (Proportion of participants reporting pain freedom at two hours post-dose)

SECONDARY OUTCOMES:
Most bothersome migraine-associated symptom | 11 weeks
  Migraine-associated symptoms: nausea, vomiting, photophobia or phonophobia and phonophobia (frequency)

CONTACTS AND LOCATIONS:
Locations (2):
- Brazil (2):
  - Eurofarma Laboratorios S.A, São Paulo, São Paulo
  - CEPIC, São Paulo, São Paulo

IPD SHARING:
Plan to Share IPD: No